CLINICAL TRIAL: NCT03932591
Title: The Effect of Inhibitory Kinesio Taping Application on Severity of Spasticity, Increased Stretch Reflex and Motor Neuron Activity: Prospective, Randomized, Controlled Trials
Brief Title: The Effect of Inhibitory Kinesio Taping Application on Spasticity, Stretch Reflex and Motor Neuron Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstPMRTRH-KT1
Record Dates: First submitted 2019-04-28; First posted 2019-04-30 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Muscle Physiology
Keywords: Spasticity; kinesio tape; stretch reflex; H-reflex; T-reflex
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: intervention group: inhibitory kinesio taping application in spastic hemiplegic patients controlled group: sham kinesio taping application in spastic hemiplegic patients
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Inhibitory kinesio taping method will be used for intervention group. Y shaped, 34-40 cm length, 5 cm width, skin color kinesio tape will be applied on spastic gastrocsoleus muscle. The base of Y shaped tape will be strapped on calcaneus ( no stretch for first 5 cm) and the both legs of Y shaped tape will be strapped on gastrocnemius muscle medial and lateral head with 15% stretch.
  Interventions: Procedure: kinesio taping method
- Control (Sham Comparator): Sham kinesio tape will be used for controlled group. 2,5 cm width, 5 cm length, skin color 2 pieces kinesio tape will be applied on medial and lateral head of gastrocnemius muscle without stretch. 5 cm length, 5 cm width, skin color 1 piece kinesio tape will be applied on achilles tendon without stretch.
  Interventions: Procedure: Sham kinesio taping

INTERVENTIONS:
Procedure: kinesio taping method — Kinesio tape is an elastic, adhesive, hypo-allergenic, latex-free tape. Kinesio taping method is rehabilitative taping technique. One of the purposes of this technique is to facilitate or inhibit the muscles.
  Other Names: Antispastic modality
  Arms: intervention
Procedure: Sham kinesio taping — Sham kinesio tape will be used for controlled group. 2,5 cm width, 5 cm length, skin color 2 pieces kinesio tape will be applied on medial and lateral head of gastrocnemius muscle without stretch. 5 cm length, 5 cm width, skin color 1 piece kinesio tape will be a
  Other Names: Sham antispastic application
  Arms: Control

SUMMARY:
The first aim of this study is whether the inhibitory kinesio taping application can reduce spasticity. The second aim of this study is to investigate whether the kinesio taping application have neuromodulatory activity on motor neuron and stretch reflex.

Hypotheses of this study: unlike healthy cases, in patients with spastic hemiplegia

1. Inhibitory kinesio taping application can reduced spasticity
2. Inhibitory kinesio taping application can reduced motor neuron activity and stretch reflex

DETAILED DESCRIPTION:
This study will include 78 spastic hemiplegic patient ( 39 controlled, 39 intervention group) Spasticity , Soleus Hmax/Mmax, Soleus T reflex, Soleus H reflex will be evaluated in this study.

Inhibitory kinesio taping method will be used in intervention group for 64-66 hours. Y shaped kinesio tape will be applied on spastic gastrocsoleus muscle. Sham kinesio taping method will be used in controlled group for 64-66 hours. 2 pieces kinesio tape 2,5 cm width, 5 cm length will be applied on gastrocnemius medial and lateral head, 1 piece kinesio tape 5 cm width, 5 cm length will be applied on achilles tendon.

Spasticity, Soleus Hmax/Mmax, Soleus T reflex and H reflex will be measured pre-application (T0), after-application ( in a few minutes) (T1), after 64-66 hours ( with band applied) (T2) and after band removed (T3). Spasticity in both groups will be evaluated with modified ashworth scale.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ischemic/hemorrhagic stroke
* First stroke attack
* Gastrocsoleus muscle spasticity ( Modified Ashworth Scale 1-3)

Exclusion Criteria:

* Perform surgery from the related limb
* Skin problems, wounds and infections
* Allergy to the kinesio tape material
* Antispastic drug use
* Contracture in gastrocsoleus muscle or antagonists
* Peripheral nerve lesion in the lower extremity
* II.Motor neuron diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 72 hours
  Muscle tone measure. Range 0 (No increase in muscle tone) to 4 (Affected part(s) rigid in flexion or extension)

SECONDARY OUTCOMES:
Hmax/Mmax rate | 72 hours
  Motor neuron activity will be determined by using the Hmax/Mmax rate. A higher rate indicates higher motor neuron activity.
T-reflex amplitude | 72 hours
  The stretch reflex activity will be evaluated by using T-reflex amplitude. The unit of this variable is microvolts. A higher amplitude indicates higher stretch reflex activity.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Ekici Zincirci, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li S, Francisco GE. New insights into the pathophysiology of post-stroke spasticity. Front Hum Neurosci. 2015 Apr 10;9:192. doi: 10.3389/fnhum.2015.00192. eCollection 2015. PMID 25914638
- [Background] Qafarizadeh F, Kalantari M, Ansari NN, Baghban AA, Jamebozorgi A. The effect of kinesiotaping on hand function in stroke patients: A pilot study. J Bodyw Mov Ther. 2018 Jul;22(3):829-831. doi: 10.1016/j.jbmt.2017.09.015. Epub 2017 Sep 23. PMID 30100319
- [Background] Karadag-Saygi E, Cubukcu-Aydoseli K, Kablan N, Ofluoglu D. The role of kinesiotaping combined with botulinum toxin to reduce plantar flexors spasticity after stroke. Top Stroke Rehabil. 2010 Jul-Aug;17(4):318-22. doi: 10.1310/tsr1704-318. PMID 20826420
- [Background] Tamburella F, Scivoletto G, Molinari M. Somatosensory inputs by application of KinesioTaping: effects on spasticity, balance, and gait in chronic spinal cord injury. Front Hum Neurosci. 2014 May 30;8:367. doi: 10.3389/fnhum.2014.00367. eCollection 2014. PMID 24910607
- [Background] Alexander CM, McMullan M, Harrison PJ. What is the effect of taping along or across a muscle on motoneurone excitability? A study using triceps surae. Man Ther. 2008 Feb;13(1):57-62. doi: 10.1016/j.math.2006.08.003. Epub 2006 Dec 22. PMID 17188548
- [Background] Yoosefinejad AK, Motealleh A, Abbasalipur S, Shahroei M, Sobhani S. Can inhibitory and facilitatory kinesiotaping techniques affect motor neuron excitability? A randomized cross-over trial. J Bodyw Mov Ther. 2017 Apr;21(2):234-239. doi: 10.1016/j.jbmt.2016.06.011. Epub 2016 Jun 17. PMID 28532863